CLINICAL TRIAL: NCT03870074
Title: Cardiopulmonary Exercise Test Predicts Long-term Survival and Positive Response to Cardiac Resynchronization Therapy.
Brief Title: CPET Predicts Long-term Survival and Positive Response to CRT
Acronym: CPET-CRT
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: 2.30/IV/09
Record Dates: First submitted 2019-02-21; First posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: heart failure; cardiac resynchronization therapy; cardiopulmonary exercise test; responders to CRT; non-responders to CRT; survival prognosis after CRT
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responders: Patients with improvement of at least one NYHA class after one year from CRT.
- Non-responders: Patients with no improvement of at least one NYHA class after one year from CRT.

SUMMARY:
The study tested the usefulness of cardiopulmonary exercise test (CPET) in selection of potential responders to CRT.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) is an acknowledged therapy of selected patients with heart failure (HF). One of the unresolved problems is high percentage of non-responders to CRT, reaching 40%. No single parameter, helpful in identifying non-responders prior to CRT implantation, was found.

The study included patients with HF of ischemic or non-ischemic etiology, in NYHA class II-IV, EF≤35% and QRS≥120ms. All the patients had CRT implanted. Clinical evaluation, CPET and NT-proBNP levels measurement were performed before CRT implantation and after 3-6 months. Improvement in HF symptoms of one or more NYHA class correlated with two-years survival. It was used as the criterion of positive response to CRT.

ELIGIBILITY:
Inclusion Criteria:

* HF in class III or IV according to New York Heart Association (NYHA) in the course of ischemic (ICM) or non-ischemic cardiomyopathy (NICM), QRS complex duration ≥ 120ms, EF ≤35% and dilatation of the left ventricle diastolic diameter >55mm (LVdD), according to the ESC guidelines in 2007
* HF in NYHA class II, LBBB with QRS complex duration ≥ 150 ms according to the guidelines update in 2010
* optimal pharmacotherapy of HF in the period of three months prior to the study entry.
* the expected survival of the patient > 1 year.

Exclusion Criteria:

* severe chronic obstructive pulmonary disease (FEV1 <30%)
* inability to perform a stress test on a treadmill

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study comprised 122 patients qualified for CRT-D and followed-up for five years after CRT implantation. Patients were qualified for CRT-D based on the guidelines of the European Society of Cardiology in 2007 and its update in 2010.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Death | Follow up within 5 years from CRT
  All cause death, data from hospital entries and phone follow-up .
Heart transplantation | Follow up within 5 years from CRT
  Heart transplantation as the definitive therapy of end-stage heart failure.

SECONDARY OUTCOMES:
Positive response to CRT | Follow up within 1 year from CRT
  Positive response to CRT was defined as the improvement in heart failure symptoms of 1 or more NYHA classes

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Chwyczko, MD,PhD, Principal Investigator — Institute of Cardiology

IPD SHARING:
Plan to Share IPD: No